CLINICAL TRIAL: NCT06367777
Title: Investigating the Effects of the Neuromodulation of the Cervical and the Low-thoracic Spinal Cord on Nociceptive Processing in Healthy Volunteers - an Randomized, Sham-controlled, Double-blinded Study
Brief Title: Cervical/Thoracic Neuromodulation and Nociceptive Processing
Acronym: MICROVOLT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024/14MAR/132
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Nociceptive Pain
Keywords: tsDCS; non-invasive neuromodulation; healthy volunteers
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal cervical tsDCS (Experimental): Participants will receive:
  1. 20 minutes of 2.5 milliamperes (mA) anodal tsDCS at the cervical level.
  2. 20 minutes of sham tsDCS at the low-thoracic level.
  Interventions: Device: cervical a-tsDCS
- Anodal thoracic tsDCS (Experimental): Participants will receive:
  1. 20 minutes of sham tsDCS at the cervical level.
  2. 20 minutes of 2.5 milliamperes (mA) anodal tsDCS at the low-thoracic level.
  Interventions: Device: thoracic a-tsDCS
- Sham tsDCS (Sham Comparator): Participants will receive:
  1. 20 minutes of sham tsDCS at the cervical level.
  2. 20 minutes of sham tsDCS at the low-thoracic level.
  Interventions: Device: sham tsDCS

INTERVENTIONS:
Device: cervical a-tsDCS — Anodal transcutaneous spinal direct current stimulation (a-tsDCS)
  Arms: Anodal cervical tsDCS
Device: thoracic a-tsDCS — Anodal transcutaneous spinal direct current stimulation (a-tsDCS)
  Arms: Anodal thoracic tsDCS
Device: sham tsDCS — Sham transcutaneous spinal direct current stimulation (s-tsDCS)
  Arms: Sham tsDCS

SUMMARY:
Several studies have demonstrated that direct currents delivered through the skin at the level of the low-thoracic spinal cord can influence spinal cord function. In human volunteers, anodal low-thoracic transcutaneous spinal direct current stimulation (tsDCS) alters spinal processing of nociceptive inputs. Whether cervical tsDCS is able to do the same is less well known. In this double-blinded, sham-controlled and cross-over trial, the investigators will compare the effects on the nociceptive processing of healthy volunteers of cervical and low-thoracic tsDCS.

DETAILED DESCRIPTION:
The investigators will compare the effects on the nociceptive processing of healthy volunteers of cervical and low-thoracic tsDCS. This study will be a double-blinded, sham-controlled, cross-over trial. Each participant will undergo three experimental sessions (anodal cervical tsDCS and sham thoracic tsDCS vs. sham cervical tsDCS and anodal thoracic tsDCS vs. sham cervical tsDCS and sham thoracic tsDCS), separated by at least one week.

ELIGIBILITY:
Inclusion Criteria:

Healthy young adults

Exclusion Criteria:

* Known medical conditions (e.g., diabetes, neuropathy, psychiatric disorders, seizure, migraine, pacemaker or other implanted medical devices...)
* Use of any medication (except contraception)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in contact-heat evoked potentials amplitude | Throughout the entire study, approximately during 6 months
  N2 amplitude

SECONDARY OUTCOMES:
Change in intensity of perception to contact-heat nociceptive stimuli | Throughout the entire study, approximately during 6 months
  Numerical rating scale (0-100)
Change in skin temperature | Throughout the entire study, approximately during 6 months
  Temperature (°C)
Change in cutaneous blood flow | Throughout the entire study, approximately during 6 months
  LDF flow (PU)

CONTACTS AND LOCATIONS:
Overall Officials: André Mouraux, MD, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lenoir C, Jankovski A, Mouraux A. Anodal Transcutaneous Spinal Direct Current Stimulation (tsDCS) Selectively Inhibits the Synaptic Efficacy of Nociceptive Transmission at Spinal Cord Level. Neuroscience. 2018 Nov 21;393:150-163. doi: 10.1016/j.neuroscience.2018.10.007. Epub 2018 Oct 12. PMID 30321585
- See also: NOCIONS lab website — https://www.nocions.org